CLINICAL TRIAL: NCT05362851
Title: a Multicenter, Double-blind, Randomized, Active Drug Control, Parallel Design Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of YYC301 in Patients With Osteoarthritis of the Knee Joint
Brief Title: Clinical Trial of YYC301 P3 for Treatment of Osteoarthritis of the Knee
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yooyoung Pharmaceutical Co., Ltd. (Industry)
Collaborators: CliPSBnC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YYPCT_YYC301_301
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Celecoxib

STUDY DESIGN:
Intervention Model Description: The purpose of this study is to investigate the efficacy and safety after administration of YYC301(Experimental) or Celecoxib(Comparator) in subjects with knee osteoarthritis in a state of uncontrolled pain who took Celecoxib(Cox-2 inhibitor).
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YYC301-1, YYC301-2, YYC301-3 & Celecoxib placebo (Experimental): * YYC301-1 is a capsule. It is composed of Celecoxib 200mg and Tramadol 37.5mg complex.
  * YYC301-2 is a capsule. It is composed of Celecoxib 200mg and Tramadol 75mg complex.
  * YYC301-3 is a capsule. It is composed of Celecoxib 200mg and Tramadol 150mg complex.
  Interventions: Drug: YYC301-1 & YYC301-2 & YYC301-3
- YYC301-1 placebo, YYC301-2 placebo, YYC301-3 placebo & Celecoxib (Active Comparator): Concomitant Drugs with Celecoxib 200mg and YYC301-1 placebo one capsule.
  Concomitant Drugs with Celecoxib 200mg and YYC301-2 placebo one capsule.
  Concomitant Drugs with Celecoxib 200mg and YYC301-3 placebo one capsule.
  Interventions: Drug: YYC301 placebo & Celecoxib 200mg

INTERVENTIONS:
Drug: YYC301-1 & YYC301-2 & YYC301-3 — YYC301-1: Subjects take the investigational products once a day
  YYC301-2: Subjects take the investigational products once a day
  YYC301-3: Subjects take the investigational products once a day
  Other Names: YYC301-1: Tramadol 37.5Mg+ Celecoxib 200mg; YYC301-2: Tramadol 75mg+ Celecoxib 200mg; YYC301-3: Tramadol 150mg+ Celecoxib 200mg
  Arms: YYC301-1, YYC301-2, YYC301-3 & Celecoxib placebo
Drug: YYC301 placebo & Celecoxib 200mg — comparator medication
  Arms: YYC301-1 placebo, YYC301-2 placebo, YYC301-3 placebo & Celecoxib

SUMMARY:
A Multi-center, Double-blinded, Randomized, Active-controlled, Parallel Design, phase 3 Clinical Trial to Evaluate the Efficacy and Safety of YYC301 in Patients with Osteoarthritis of the Knee Joint

ELIGIBILITY:
Inclusion Criteria:

* Men/Women aged over 20
* Subjects who are diagnosed with one- or both-sided knee osteoarthritis according to the standards of clinical diagnosis from American College of Rheumatology(ACR)have knee osteoarthritis pain and meet over three of the following conditions.

  1. Older than 50
  2. Morning stiffness for less than 30 minutes
  3. Crepitus on active motion
  4. Bony tenderness
  5. Bony enlargement
  6. Not have heat-generating site
* Subjects who are diagnosed with degenerative osteoarthritis and have its pain at least for over 3 months before the screening visit.
* Subjects who are uncontrolled with pain after administration of Celecoxib at least for over 2 weeks before the randomization and have more than 50mm out of 100mm VAS at randomization.
* Subjects who voluntarily agree to participate in this clinical trial in writing.

Exclusion Criteria:

* Subjects with rheumatoid arthritis or inflammatory, infectiousand metabolic arthritis.
* Subjects with ochronosis, hemochromatosis, secondary knee osteoarthritis by systemic disease.
* Subjects who have severe pain such as Sudek's atrophy, Paget's disease and spinal disc herniation.
* Subjects with poly-articular affected by severe pain of knee osteoarthritis.
* Subjects who take psychtrophic medicine and narcotic analgesics for over 3 months that might affect on pain sensory system.
* Subjects who had Tramadol but there was no improvement in pain.
* Subjects who got the follwing treatment and medicine before the screening;

  1. Subjects who had surgery on knee ligaments within a year, cartilage transplant and scarf osteotomy.
  2. Subjects who had arthroscopy within 6 months.
  3. Subjects with intra-articular knee joint steroid injection within 3 months.
  4. Subjects with HA injection in knee joint within 6 months.
  5. Subjects with systemic steroid injection within a month(but inhaled steroids)
  6. Subjects with knee replacement surgery.
* Subjects who hot the following treatment and medicine before the randomization;

  1. Subjects who had Celecoxib, acetaminophen or steroidal/non-steroidal anti-inflammatory drugs except low dose aspirin(before 300mg/day) But, acetaminophen and low dose aspirin (before 300mg/day) are prohibited within 24 hours)
  2. Nutritional supplements, physical therapy and Korean herbal medicine for knee osteoarthritis and it pain within 2 weeks.
* Subjects who have to take anticoagulant drugs such as warfarin and coumarin during this clinical trial.
* Subjects who took MAO inhibitors within 14 days before the screening or needed to take these drugs during this clinical trials.
* Subjects with drug and opioid hypersensitivity and who have history.
* Subjects with sulfanilamide allergy and who have history.
* Subjects with asthmma, acute rhinitis, nasal polyp, angioedema, urticaria, allergic reaction to aspirin or any oher NSAIDs(incluing COX-2 inhibitors)
* Subjects with significant investigations - Hyperkalemia(Exceeded 5.5mmol/L)
* Subjects with severe liver dysfunction (ALT or AST of more than 3.0 times the upper limit of ULN and 1.5 tmines the upper limit of ULN)
* Subjects with severe renal impairment (Serum Creatine > 3x ULN).
* Subjects with active peptic ulcer and gastrointestinal bleeding.
* Severe blood disease (Agranulocytosis, aplastic anemia, hemolytic anemia, Thrombocytopenia, etc.).
* Subjects with Crohn's disease or inflammatory bowel disease such as ulcerative clitis.
* Subjects with congestive heart failure(NYHA 2-4)
* Subjects with severe ischaemic heart disease, peripheral artery disease and/or cerebrovascular disease.
* Subjects with genetic problesa such as galactose intolerance), lapp lactase deficiency or glucose-galactose malabsorption).
* Subjects with acute alcohol intoxification.
* Subjects who are addicted with took central nervous system drugs such as painkillers, sleeping pills, anti-anxiety medications, etc.
* Subjects with severe bronchopulmonary dysplasia.
* Subjects with head injury history of brain structure lesions which may be in danger of mental confusion.
* Subjects with epilepsy who are treated properly.
* Subjects who use Tramadol to cure for narcotic withdrawal.
* Subjects who took other clinical drugs more than once within 30 days before the clinical trial.
* Subjects suspected to be pregnant who don't agree with the clinical method which is permitted medically during clinical trial(Method of hormone contraception, IUD(Intrauterine device) or IUS(Intrauterine system)), tubal ligation, bilateral tubal ligation(condom, Diaphragm, etc).
* Pregnant woman and breastfeeding woman.
* Subjects who can increase risk due to clinical test and administraion of drugs or have severe grade / chronic medical, mental condition or abnormal laboratory result that may interfere with the analysis of thest results.
* Any other ineligible condition at the direction of investigator that would be ineligible to participate the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
100mm Pain VAS | at 13 weeks after randomization after administration of YYC301(Experimental drug).
  Subjects who have severe pain at one-or both sided knee osteoarthritis directly assess the degree of pain (within 24 hours) with a straight line which has 0mm to 100mm. 0 mm means 'doesn't have pain' and 100 mm means 'maximum pain who can imagine'.In order to investigate the degree of subject's pain change from administration of YYC301(Experimental drug).

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Ho Yoon, Ph.D., Principal Investigator — Kyunghee University Medical Center
Locations (1):
- KyungHee University Medical Center, Seoul, Dongdaemun-gu /Kyung Hee Dae-ro 23, South Korea

IPD SHARING:
Plan to Share IPD: Undecided